CLINICAL TRIAL: NCT05821738
Title: Avapritinib in Relapsed Refractory or MRD-positive CBF-AML With KIT Mutations
Brief Title: Avapritinib in CBF-AML With KIT Mutations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Chen Suning, Principal Investigator, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZ-AML-KIT
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Core Binding Factor Acute Myeloid Leukemia; KIT Mutation-Related Tumors
MeSH Terms: interventions — avapritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental): The treatment group will receive avapritinib orally. The dosage is 100mg to 300mg qd, allowed to combine with other chemotheray drugs.
  Interventions: Drug: Avapritinib

INTERVENTIONS:
Drug: Avapritinib — administered orally

SUMMARY:
AML with t(8; 21)(q22; q22) or inv(16)(p13; q22)/t(16; 16)(p13; q22) is known as CBF-AML. KIT mutations are common in CBF-AML, which have a worse prognosis.This study is aimed to evaluate the efficacy of Avapritinib, an highly specific inhibitor of the KIT gene, in CBF-AML with KIT mutations.

DETAILED DESCRIPTION:
Acute Myeloid Leukemia (AML) with the chromosomal abnormality of t(8; 21)(q22; q22) or inv(16)(p13; q22)/t(16; 16)(p13; q22) is known as the Core Binding Factor AML (CBF-AML). KIT mutation is a common mutation in CBF-AML, which is more likely to relapse and have a worse prognosis.

Avapritinib is an oral tyrosine kinase inhibitor (TKI) with selective inhibitory activity against KIT and PDGFRA. Avapritinib has been approved by FDA for the treatment of gastrointestinal stromal tumors(GIST) with PDGFRA mutations and Advanced systemic mastocytosis (AdvSM). However, the efficacy of avapritinib in AML with KIT mutations is uncertain.

This prospective, multicenter clinical study of the efficacy and safety of avapritinib in relapsed refractory or molecular minimal residual disease (MRD)-positive AML with KIT mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute myeloid leukemia accompanied by t(8; 21)/RUNX1-RUNX1T1, or inv(16)/t(16; 16)/CBFβ-MYH11;
2. Accompanied by KIT mutation
3. Disease recurrence after the first remission, or the mol-MRD remains positive after the morphologic remission of AML.
4. No active infection.
5. Liver function: TBIL≤ 2×ULN,ALT/AST≤ 3×ULN, CCr ≥ 50ml/min，NYHA grading ≤2; SaO2 >92%.
6. ECOG <2;

(11) Predicted survival > 12 weeks.

Exclusion Criteria:

1. Accept other AML targeted therapies, such as dasatinib, sorafenib, gilteritinib, etc. simultaneously;
2. The presence of uncontrolled and active infections (including bacterial, fungal or viral infections).
3. Underlying diseases such as myocardial infarction, chronic heart failure, decompensated liver dysfunction, renal failure, etc.
4. Pregnant or lactating women;
5. Accompanied by other malignant tumors requiring treatment;
6. Other interventional clinical studies have been enrolled.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite complete remission (CRc) | Assessed at protocol-defined timepoints through end of study, up to approximately 36 months.
  The proportion of participants who achieve Composite complete remission (CRc)，which includes complete remission (CR)、CR with partial hematologic recovery (CRh)、CR with incomplete blood count recovery (CRi) and morphology leukemia free (MLFS) based on response criteria for AML.

SECONDARY OUTCOMES:
MRD-negative rate | Assessed at protocol-defined timepoints through end of study, up to approximately 36 months.
  The proportion of participants who achieve a negative molecular MRD.
Progression-free survival (PFS) | From the first day of treatment until any failure (resistant disease, relapse, or death), assessed up to 1 to 3 years.
  The Kaplan-Meier method will be used to assess PFS probabilities.
Overall survival (OS) | From the first day of treatment to time of death from any cause, assessed up 1 to 3 years.
  The Kaplan-Meier method will be used to assess OS probabilities.
Incidence of adverse events (AEs) | Up to approximately 1 to 3 years.
  Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. The proportion of patients with AEs will be estimated, along with the 95% credible interval.

CONTACTS AND LOCATIONS:
Overall Officials: Suning Chen, Principal Investigator — First Affiliated Hospital of Soochow University
Locations (1):
- First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China